CLINICAL TRIAL: NCT05477706
Title: Use of a Peer Intervention to Improve Access Among Rural Women Veterans With Psychological Distress and Unmet Social Needs
Brief Title: Peer Intervention to Improve Access Among Rural Women Veterans With Psychological Distress and Unmet Social Needs
Acronym: EMBER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Syracuse VA Medical Center (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-50334; 1652536 (Other: Syracuse VA Medical Center IRB)
Record Dates: First submitted 2022-07-06; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Psychological Distress; Depression; PTSD; Anxiety
Keywords: Peer-delivered Intervention; Psychological Distress; Unmet social needs; Rural Women Veterans; PTSD; Depression; Suicide risk; Telehealth; Anxiety
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Support for Progress (PSP) (Experimental): PSP includes an initial 60-minute video or phone appointment and then follow-up tailored to the Veteran's preferences. The Peer Specialist guides the Veteran through a card-sorting task to prioritize concerns and then create a personalized care plan. The Peer then provides up to six months of outreach and support to implement the care plan. At the end of the six months, the Veteran and peer review the plan, determine next steps and consider other supports and resources to sustain progress made.
  Interventions: Other: Personalized Support for Progress (PSP)
- Tailored Referral (TR) (Active Comparator): The Tailored Referral (TR) comparator will be comprised of written or emailed information describing resources and contact information for VHA and local social and mental health resources. Examples include information about the appropriate office/person to reach within the local VA or area, help scheduling an appointment, or information for a same-day Primary Care - Mental Health Integration (PCMHI) assessment.
  Interventions: Other: Tailored Referral (TR)

INTERVENTIONS:
Other: Personalized Support for Progress (PSP) — Personalized Support for Progress (PSP) is a Peer Specialist delivered intervention in which a peer supports Veterans in prioritizing their needs and attaining access to the Veterans' preferred services.
  Arms: Personalized Support for Progress (PSP)
Other: Tailored Referral (TR) — TR consists of detailed resource information and referral, consistent with standard practice.
  Arms: Tailored Referral (TR)

SUMMARY:
This research project will refine and evaluate delivery of a peer-delivered evidence-based intervention to improve perceived access and actual engagement with mental health treatment and social resource service use among rural women Veterans, especially Veterans of color, with psychological distress and unmet social needs.

DETAILED DESCRIPTION:
Not only do rural women Veterans report significant psychological distress (PTSD, anxiety, depression, suicide risk) and social needs (housing, transportation, material insecurity), they also experience substantial barriers accessing services which limits the Veteran Health Administration's (VHA) ability to address their needs. Personalized Support for Progress (PSP) is a virtually delivered intervention in which a Peer Specialist supports Veterans in prioritizing their needs and attaining access to the Veterans' preferred services. This trial is investigating whether PSP with rural women Veterans is associated with improved perceived access and actual engagement to mental health and social resource services, as well as high satisfaction and improved mental health, social needs and function outcomes. Rural women Veterans of color are more likely to be coping with psychological distress and social needs, as well as experiencing barriers to engagement and retention in services. Therefore this trial is designed to ensure that PSP delivery is tailored to increase rural women Veterans of color's acceptability.

The primary study design is a randomized controlled trial of Tailored Referral Information (TR) compared to Personalized Support for Progress (PSP) intervention for rural women Veterans with psychological distress and social needs (Aim 2). Prior to implementing the trial, focus groups and individual interviews will be conducted with women Veterans, Peer Specialists, and providers/stakeholders to determine any needed adaptations to determine any needed adaptations of PSP delivery for rural women Veterans and for PSP implementation in rural primary care clinics (Aim 1).

ELIGIBILITY:
Aim 1 (Focus groups and interviews with women Veterans, Peer Specialists, and Providers to assess adaptations needed for PSP prior to the intervention trial)

Inclusion Criteria:

Veteran Inclusion:

* Veteran status (non-Veterans will not be enrolled in this trial)
* Identifies as a woman or as gender fluid
* Resides in a rural or highly rural area
* Psychological distress in the past 6 months as evidenced by a diagnosis in the electronic health record or elevated score on the PHQ-9, GAD-7 and/or PCL
* At least one social need in the past 6 months on the PRAPARE
* Ability to communicate in English including reading, writing, hearing, and speaking well enough to complete research and intervention tasks.

Providers Inclusion Criteria:

• Any provider (physician, social worker, therapist, etc. with experience working with rural women Veterans) employed by the VHA

Peers inclusion criteria:

•Any peer specialist employed by the VHA who identifies as a woman or as gender fluid

Veteran Exclusion Criteria:

* Any Veteran with high suicide or homicide risk and/or evaluated by the PI or another clinician to be clinically unstable
* Veterans with impairment that would not allow them to engage in study activities including active psychosis, cognitive deficits, severe substance use requiring detoxification (documented in electronic health record or reported by a primary care clinician team member)

Aim 2 (Randomized controlled trial of PSP compared to TR)

Inclusion:

* Veteran status (non-Veterans will not be enrolled in this trial)
* Identifies as a woman or as gender fluid
* Resides in a rural or highly rural area
* Veteran must reside in Southeastern Texas, Arkansas or Louisiana
* Psychological distress in the past 6 months as evidenced by a diagnosis in the electronic health record or elevated score on the PHQ-9, GAD-7 and/or PCL
* At least one social need in the past 6 months on the PRAPARE
* Ability to communicate in English including reading, writing, hearing, and speaking well enough to complete research and intervention tasks.

Exclusion:

* Any Veteran with high suicide or homicide risk and/or evaluated by the PI or another clinician to be clinically unstable
* Veterans with impairment that would not allow them to engage in study activities including active psychosis, cognitive deficits, severe substance use requiring detoxification (documented in EMR or reported by a PACT member)
* Veterans who have current VA or non-VA peer support engagement (an appointment within the last month and/or additional follow-up scheduled)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identification as woman or gender fluid
Enrollment: 72 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in actual engagement with social resource services and mental health treatment | Baseline, 6 Months (post-intervention), and 9 Months (3 Months post-intervention)
  VHA Administrative data will be used to assess face-to-face and digital visits (encounters) along with self-reported number of visits on the Epidemiological Catchment Area Survey (ECA).
Change in perceived access to social resource services and mental health treatment | Baseline, 6 Months (post-intervention), and 9 Months (3 Months post-intervention)
  The Assessment of Perceived Access to Care (APAC) measure will be used to assess perceived access to social resource services and mental health treatment at each time-point with a scale of 1-5 so that higher total scores equals better access.

SECONDARY OUTCOMES:
Veteran satisfaction | 6 Months (post-intervention) and 9 Months (3 Months post-intervention)
  Veteran satisfaction will be measures using the Client Satisfaction Questionnaire-8 (CSQ-8), an 8 item measure of participant satisfaction with services. An overall score is calculated by summing the respondent's rating (item rating) score for each scale item. For the CSQ-8 scores range from 8 to 32, with higher values indicating higher satisfaction.
Change in depression symptoms | Baseline, 6 Months (post-intervention), and 9 Months (3 Months post-intervention)
  Change in depression symptoms for Veteran participants will be assessed using the Patient Health Questionnaire (PHQ)-9, a self-administered depression scale. The total score can range from 1 to 27 with a higher score indicating more severe depression.
Change in social needs | Baseline, 6 Months (post-intervention), and 9 Months (3 Months post-intervention)
  Change in social needs will be assessed using the Protocol for Responding to and Assessing Patients' Assets, Risks, and Experiences (PRAPARE), a standardized tool for collecting social determinants of health (SDH) data including socioeconomic and psychosocial characteristics. The total score can range from 0 to 22 with the total cumulative score indicating presence of risk and unmet needs.
Change in greater perceived progress on needs | Baseline, 6 Months (post-intervention), and 9 Months (3 Months post-intervention)
  An adapted version of the Goal Attainment Scale (GAS) will be used to assess Veteran perceived progress on needs. The GAS is a functional scale used to measure the extent of progress towards individual goals during the course of an intervention. Each subject has their own outcome measures but they are scored in a standardized way. Scale items are based on current and expected levels of performance.
Change in functioning | Baseline, 6 Months (post-intervention), and 9 Months (3 Months post-intervention)
  The Brief Inventory of Psychosocial Functioning (B-IPF) will be used to measure change in functioning. The B-IPF is an 7-item self-report instrument measuring PTSD-related functional impairment in the past 30 days by looking at seven functional domains including romantic relationships, family relationships, work, friendships and socializing, parenting, education, and self-care. Items are scored on a Likert scale from 0 to 6. The B-IPF is scored by summing the scored items to create a total score, dividing the total score by the maximum possible score based on the number of items scored, and multiplying by 100. The B-IPF represents an overall index of functioning, with higher scores indicating greater functional impairment.
Change in Perception of Quality of Life | Baseline, 6 Months (post-intervention), and 9 Months (3 Months post-intervention)
  The World Health Organization Quality of Life (WHO-QOL) measure will be used to assess quality of life (QOL) for each participant in the context of culture, value systems, personal goals, standards and concerns. The scale is scored between 0 to 100 with higher scores indicating a higher quality of life.
Stigma-related beliefs about mental health | Baseline, 6 Months (post-intervention), and 9 Months (3 Months post-intervention)
  The Endorsed and Anticipated Stigma Inventory (EASI) is a tool for assessing beliefs about mental illness and mental health treatment among Veterans. The scales are scored so that higher scores are indicative of greater stigma.
Change in perceived stress | Baseline, 6 Months (post-intervention), and 9 Months (3 Months post-intervention)
  The Perceived Stress Scale (PSS) will be used to measure each participants subjective understanding of their psychological stress level in the past month. Scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Change in anxiety symptoms | Baseline, 6 Months (post-intervention), and 9 Months (3 Months post-intervention)
  Change in anxiety symptoms for Veteran participants will be assessed using the Generalized Anxiety Disorder (GAD)-7, a seven-item instrument used to measure the severity of generalized anxiety disorder (GAD). The total score can range from 0 to 21 with a higher score indicating a larger amount of anxiety symptoms.
Change in Post-Traumatic Stress Disorder (PTSD) symptoms | Baseline, 6 Months (post-intervention), and 9 Months (3 Months post-intervention)
  Change in PTSD symptoms for Veteran participants will be assessed using the Post Traumatic Stress Disorder (PTSD) Checklist (PCL-5), a 20-item self-report measure that assesses the 20 Diagnostic and Statistical Manual-5 symptoms of PTSD. For this trial a score of 31 or higher indicates a positive screen for PTSD.

OTHER OUTCOMES:
Therapeutic alliance | Baseline, 6 Months (post-intervention), and 9 Months (3 Months post-intervention)
  The Kim Alliance Scale (KAS-R) will be used to assess the quality of the therapeutic alliance between the Veteran and provider along with patient empowerment and satisfaction with the relationship.
Perceived Confidence | Baseline, 6 Months (post-intervention), and 9 Months (3 Months post-intervention)
  The Perceived Confidence Scale will be used to assess each participants' feelings of confidence in engaging in tasks independently.
Autonomy Support | Baseline, 6 Months (post-intervention), and 9 Months (3 Months post-intervention)
  The Autonomy Support Questionnaire will be used to assess each participants perceptions of autonomy support from their provider or peer.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Poleshuck, PhD, Principal Investigator — Syracuse VA Medical Center; Derrecka Boykin, PhD, Principal Investigator — Michael E. DeBakey Medical Center
Locations (2):
- United States (2):
  - Syracuse VA Medical Center, Syracuse, New York
  - Michael E. DeBakey VA Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Once all data collection is complete and the coded database is finalized, individual participant data (IPD) will be shared according to PI discretion. For instance, IPD may be shared to be used in meta-analyses or other review papers. No identifiable participant information will be shared.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data will be available once the database is finalized and will remain available in the future.
Access Criteria: Access to the data can be obtained by emailing the PIs and describing the reason the data is needed.

REFERENCES:
- [Background] Fortney JC, Pyne JM, Hawrilenko M, Bechtel JM, Moore D, Nolan JP, Pfeiffer P, Shushan S, Shore JH, Bowen D. Psychometric Properties of the Assessment of Perceived Access to Care (APAC) Instrument. J Ambul Care Manage. 2021 Jan/Mar;44(1):31-45. doi: 10.1097/JAC.0000000000000358. PMID 33165120
- [Background] Moreau JL, Cordasco KM, Young AS, Oishi SM, Rose DE, Canelo I, Yano EM, Haskell SG, Hamilton AB. The Use of Telemental Health to Meet the Mental Health Needs of Women Using Department of Veterans Affairs Services. Womens Health Issues. 2018 Mar-Apr;28(2):181-187. doi: 10.1016/j.whi.2017.12.005. Epub 2018 Jan 12. PMID 29339013
- [Background] Cordasco KM, Mengeling MA, Yano EM, Washington DL. Health and Health Care Access of Rural Women Veterans: Findings From the National Survey of Women Veterans. J Rural Health. 2016 Sep;32(4):397-406. doi: 10.1111/jrh.12197. Epub 2016 Jul 28. PMID 27466970
- [Background] McCarthy JF, Blow FC, Ignacio RV, Ilgen MA, Austin KL, Valenstein M. Suicide among patients in the Veterans Affairs health system: rural-urban differences in rates, risks, and methods. Am J Public Health. 2012 Mar;102 Suppl 1(Suppl 1):S111-7. doi: 10.2105/AJPH.2011.300463. Epub 2012 Jan 25. PMID 22390583
- [Background] Thomas KH, McDaniel, J.T., Haring, E.L., Albright, D.L., Fletcher, K.L. Mental health needs of military and veteran women: An assessment conducted by the Service Women's Action Network. Traumatology. 2018;24(2):104-112.
- [Background] Thomas KH, Turner, L.W., Kaufman, E.M., Paschal, A., Knowlden, A.P., Birch, D.A., Leeper, J.D. Predictors of Depression Diagnoses and Symptoms in Veterans: Results From a National Survey. Military Behavioral Health. 2015;3(4):255-265.
- [Background] Tsai J, Kasprow WJ, Kane V, Rosenheck RA. National comparison of literally homeless male and female VA service users: entry characteristics, clinical needs, and service patterns. Womens Health Issues. 2014 Jan-Feb;24(1):e29-35. doi: 10.1016/j.whi.2013.09.007. Epub 2013 Dec 15. PMID 24342077
- [Background] Brooks E, Novins DK, Thomas D, Jiang L, Nagamoto HT, Dailey N, Bair B, Shore JH. Personal characteristics affecting veterans' use of services for posttraumatic stress disorder. Psychiatr Serv. 2012 Sep 1;63(9):862-7. doi: 10.1176/appi.ps.201100444. PMID 22707088
- [Background] Renteria-Szelwach C, Steinkogler, J., Badger, E.R., & Muttukumaru, R. Transitioning to the Civilian Workforce: Issues Impacting the Reentry of Rural Women Veterans. Journal of Rural Social Sciences. 2011;26(3).
- [Background] Lehavot K, Beckman KL, Chen JA, Simpson TL, Williams EC. Race/Ethnicity and Sexual Orientation Disparities in Mental Health, Sexism, and Social Support among Women Veterans. Psychol Sex Orientat Gend Divers. 2019;6(3):347-358. doi: 10.1037/sgd0000333. PMID 31435497
- [Background] Montgomery AE, Tsai J, Blosnich JR. Demographic Correlates of Veterans' Adverse Social Determinants of Health. Am J Prev Med. 2020 Dec;59(6):828-836. doi: 10.1016/j.amepre.2020.05.024. Epub 2020 Nov 18. PMID 33220754
- [Background] Montgomery AE, Szymkowiak, D., & Tsai, J. Housing Instability and Homeless Program Use Among Veterans: The Intersection of Race, Sex, and Homelessness. Housing Policy Debate. 2020;30(3):396-408.
- [Background] Spoont M, Nelson D, van Ryn M, Alegria M. Racial and Ethnic Variation in Perceptions of VA Mental Health Providers are Associated With Treatment Retention Among Veterans With PTSD. Med Care. 2017 Sep;55 Suppl 9 Suppl 2:S33-S42. doi: 10.1097/MLR.0000000000000755. PMID 28806364
- [Background] Brooks E, Dailey N, Bair B, Shore J. Rural women veterans demographic report: defining VA users' health and health care access in rural areas. J Rural Health. 2014 Spring;30(2):146-52. doi: 10.1111/jrh.12037. Epub 2013 Jul 19. PMID 24689540
- [Background] Washington DL, Bean-Mayberry B, Riopelle D, Yano EM. Access to care for women veterans: delayed healthcare and unmet need. J Gen Intern Med. 2011 Nov;26 Suppl 2(Suppl 2):655-61. doi: 10.1007/s11606-011-1772-z. PMID 21989618
- [Background] Fortney JC, Burgess JF Jr, Bosworth HB, Booth BM, Kaboli PJ. A re-conceptualization of access for 21st century healthcare. J Gen Intern Med. 2011 Nov;26 Suppl 2(Suppl 2):639-47. doi: 10.1007/s11606-011-1806-6. PMID 21989616
- [Background] Evans EA, Tennenbaum, D.L., Washington, D.L., & Hamilton, A.B. Why Women Veterans Do Not Use VA-Provided Health and Social Services: Implications for Health Care Design and Delivery. Journal of Humanistic Psychology. 2019.
- [Background] Allicock M, Haynes-Maslow L, Johnson LS, Carpenter WR, Vines AI, Belle DG, Phillips R, Cherry MW. Peer Connect for African American breast cancer survivors and caregivers: a train-the-trainer approach for peer support. Transl Behav Med. 2017 Sep;7(3):495-505. doi: 10.1007/s13142-017-0490-4. PMID 28425087
- [Background] Chinman M, George P, Dougherty RH, Daniels AS, Ghose SS, Swift A, Delphin-Rittmon ME. Peer support services for individuals with serious mental illnesses: assessing the evidence. Psychiatr Serv. 2014 Apr 1;65(4):429-41. doi: 10.1176/appi.ps.201300244. PMID 24549400
- [Background] Wagner C, Dichter ME, Mattocks K. Women Veterans' Pathways to and Perspectives on Veterans Affairs Health Care. Womens Health Issues. 2015 Nov-Dec;25(6):658-65. doi: 10.1016/j.whi.2015.06.009. Epub 2015 Sep 1. PMID 26341566
- [Background] Kimerling R, Bastian LA, Bean-Mayberry BA, Bucossi MM, Carney DV, Goldstein KM, Phibbs CS, Pomernacki A, Sadler AG, Yano EM, Frayne SM. Patient-centered mental health care for female veterans. Psychiatr Serv. 2015 Feb 1;66(2):155-62. doi: 10.1176/appi.ps.201300551. Epub 2014 Nov 17. PMID 25642611
- [Background] Mattocks K, Casares J, Brown A, Bean-Mayberry B, Goldstein KM, Driscoll M, Haskell S, Bastian L, Brandt C. Women Veterans' Experiences with Perceived Gender Bias in U.S. Department of Veterans Affairs Specialty Care. Womens Health Issues. 2020 Mar-Apr;30(2):113-119. doi: 10.1016/j.whi.2019.10.003. Epub 2019 Nov 14. PMID 31735581
- [Background] Mattocks KM, Baldor R, Bean-Mayberry B, Cucciare M, Gerber MR, Goldstein KM, Hammer KD, Hill EE, Kroll-Desrosiers A, Prochazka AV, Sadler AG, Bastian L. Factors Impacting Perceived Access to Early Prenatal Care among Pregnant Veterans Enrolled in the Department of Veterans Affairs. Womens Health Issues. 2019 Jan-Feb;29(1):56-63. doi: 10.1016/j.whi.2018.10.001. Epub 2018 Nov 13. PMID 30446330
- [Background] Poleshuck E, Wittink M, Crean H, Gellasch T, Sandler M, Bell E, Juskiewicz I, Cerulli C. Using patient engagement in the design and rationale of a trial for women with depression in obstetrics and gynecology practices. Contemp Clin Trials. 2015 Jul;43:83-92. doi: 10.1016/j.cct.2015.04.010. Epub 2015 Apr 30. PMID 25937505
- [Background] Poleshuck E, Wittink M, Crean HF, Juskiewicz I, Bell E, Harrington A, Cerulli C. A Comparative Effectiveness Trial of Two Patient-Centered Interventions for Women with Unmet Social Needs: Personalized Support for Progress and Enhanced Screening and Referral. J Womens Health (Larchmt). 2020 Feb;29(2):242-252. doi: 10.1089/jwh.2018.7640. Epub 2019 Sep 9. PMID 31502906
- [Background] Johnson E, Possemato, K., Funderburk, J., Poleshuck, E. Pilot Trail of Personalized Support for Progress in a VA Women's Wellness Clinic. In preparation.
- [Background] Racial and Ethnic Minority Veterans. 2020. https://www.va.gov/HEALTHEQUITY/Race_Ethnicity.asp.
- [Background] U.S. Department of Health and Human Services NIoMH. Epidemiologic Catchment Area (ECA) Survey of Mental Disorders, Wave 1 (Household), 1980-1985: United States. Rockville, MD: U.S. Dept. of Health and Human Services, National Institute of Mental Health. Published 1985. Accessed.
- [Background] Attkisson CC GT, Maruish M. The client satisfaction questionnaire-8 and the service satisfaction questionnaire-30. The use of psychological testing for treatment planning and outcome assessment. American Psychological Association https://psycnet.apa.org/record/1994-97261-016. Published 1994. Accessed.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Weathers FW, Litz, B.T., Keane, T.M., Palmieri, P.A., Marx, B.P., & Schnurr, P.P. The PTSD Checklist for DSM-5 (PCL-5). 2013.
- [Background] National Association of Community Health Centers AoAPCHO, Oregon Primary Care Association, Institute for Alternative Futures. . Accelerating Strategies to Address the Social Determinants of health: Protocol for Responding to and Assessing Patients' Assets, Risks, and Experiences http://www.nachc.com/client//PRAPARE_Abstract_Tool_April_2016.pdf. Published 2016. Accessed.
- [Background] Tabak NT, Link, P.C., Holden, J., & Granholm, E. Goal Attainment scaling: Tracking goal achievement in consumers with serious mental illness. American Journal of Psychiatric Rehabilitation. 2015;18(2):173-186.
- [Background] Kleiman SE, Bovin MJ, Black SK, Rodriguez P, Brown LG, Brown ME, Lunney CA, Weathers FW, Schnurr PP, Spira J, Keane TM, Marx BP. Psychometric properties of a brief measure of posttraumatic stress disorder-related impairment: The Brief Inventory of Psychosocial Functioning. Psychol Serv. 2020 May;17(2):187-194. doi: 10.1037/ser0000306. Epub 2018 Oct 8. PMID 30299150
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of health care interventions: A theoretical framework and proposed research agenda. Br J Health Psychol. 2018 Sep;23(3):519-531. doi: 10.1111/bjhp.12295. Epub 2018 Feb 16. No abstract available. PMID 29453791
- [Background] Affairs USDoV. Rural Veterans. https://www.ruralhealth.va.gov/aboutus/ruralvets.asp. Published 2021. Accessed.
- [Background] Hamilton A. Qualitative methods in rapid turn-around health services research. Health Services Research & Development Cyberseminar. 2013.
- [Background] Morris SB. Estimating effect sizes from pretest-posttest-control group designs. Organ Res Methods. 2008;11(2):364-386.
- [Background] Hedges LV. Distribution Theory for Glass's Estimator of Effect Size and Related Estimators. Journal of Educational Statistics. 1981;6(2).
- [Background] Morris SB. Distribution of the standardized mean change effect size for meta-analysis on repeated measures. Br J Math Stat Psychol. 2000 May;53 ( Pt 1):17-29. doi: 10.1348/000711000159150. PMID 10895520
- [Background] Julious SA, Owen RJ. Sample size calculations for clinical studies allowing for uncertainty about the variance. Pharm Stat. 2006 Jan-Mar;5(1):29-37. doi: 10.1002/pst.197. PMID 17080926
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Wittink MN, Walsh P, Yilmaz S, Mendoza M, Street RL Jr, Chapman BP, Duberstein P. Patient priorities and the doorknob phenomenon in primary care: Can technology improve disclosure of patient stressors? Patient Educ Couns. 2018 Feb;101(2):214-220. doi: 10.1016/j.pec.2017.08.004. Epub 2017 Aug 8. PMID 28844522
- [Background] Wittink MN, Yilmaz S, Walsh P, Chapman B, Duberstein P. Customized Care: An intervention to Improve Communication and health outcomes in multimorbidity. Contemp Clin Trials Commun. 2016 Dec 15;4:214-221. doi: 10.1016/j.conctc.2016.10.002. Epub 2016 Oct 11. PMID 28191546
- [Background] Williams GC, Deci EL. Activating patients for smoking cessation through physician autonomy support. Med Care. 2001 Aug;39(8):813-23. doi: 10.1097/00005650-200108000-00007. PMID 11468500
- [Background] Kim SC, Boren D, Solem SL. The Kim Alliance Scale: development and preliminary testing. Clin Nurs Res. 2001 Aug;10(3):314-31. doi: 10.1177/c10n3r7. PMID 11881945
- [Background] Kim SC, Kim S, Boren D. The quality of therapeutic alliance between patient and provider predicts general satisfaction. Mil Med. 2008 Jan;173(1):85-90. doi: 10.7205/milmed.173.1.85. PMID 18251337
- [Background] Cole S, Raju M, Barrett J, Gerrity M, Dietrich A. The MacArthur Foundation Depression Education Program for Primary Care Physicians: background and rationale. Gen Hosp Psychiatry. 2000 Sep-Oct;22(5):299-358. doi: 10.1016/s0163-8343(00)80007-9. PMID 11203035
- [Background] Devlieger I, Mayer A, Rosseel Y. Hypothesis Testing Using Factor Score Regression: A Comparison of Four Methods. Educ Psychol Meas. 2016 Oct;76(5):741-770. doi: 10.1177/0013164415607618. Epub 2015 Sep 29. PMID 29795886
- [Background] Kelcey B. A robust alternative estimator for small to moderate sample SEM: Bias-corrected factor score path analysis. Addict Behav. 2019 Jul;94:83-98. doi: 10.1016/j.addbeh.2018.10.032. Epub 2018 Oct 27. PMID 30501990
- [Background] Mackinnon DP, Lockwood CM, Williams J. Confidence Limits for the Indirect Effect: Distribution of the Product and Resampling Methods. Multivariate Behav Res. 2004 Jan 1;39(1):99. doi: 10.1207/s15327906mbr3901_4. PMID 20157642
- [Background] Shrout PE, Bolger N. Mediation in experimental and nonexperimental studies: new procedures and recommendations. Psychol Methods. 2002 Dec;7(4):422-45. PMID 12530702